CLINICAL TRIAL: NCT01990469
Title: Efficacy and Safety of Gemigliptin 50mg qd Added in Patients With Type 2 Diabetes Inadequately Controlled on Glimepiride and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-DPCL010
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: T2DM
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemigliptin (Experimental): Gemigliptin 50mg qd
  Interventions: Drug: Gemigliptin
- Placebo (Placebo Comparator): Gemigliptin placebo
  Interventions: Drug: Gemigliptin placebo

INTERVENTIONS:
Drug: Gemigliptin — DPP-4 inhibitor
  Other Names: Zemiglo
  Arms: Gemigliptin
Drug: Gemigliptin placebo — Placebo of Gemigliptin
  Arms: Placebo

SUMMARY:
After a screening, a 2-week, single-blind placebo run-in, 174 patients will be randomized in a 1 : 1 ratio to the addition of either once-daily Gemigliptin 50 mg or placebo to ongoing stable doses of glimepiride in combination with metformin for 24 weeks.

DETAILED DESCRIPTION:
Subjects will visit the center on Week 6, 12, 18 and 24 during the entire 24-week treatment period. Total study duration will be approximately 26weeks and the subjects will be to practice exercise/diet control together.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 2 Diabetes Mellitus
2. Adults aged ≥ 19 years old
3. Patients with HbA1c 7%~11% at Visit 1

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change of HbAlc from baseline at Week 24 | 24 weeks